CLINICAL TRIAL: NCT06792903
Title: Effectiveness and Safety of CG-101 Eye Drops in the Treatment of Dry Eye Syndrome
Brief Title: CG-101 Eye Drops in the Treatment of Dry Eye Syndrome
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EyeEntFudan-CG101
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Dry Eye
Keywords: dry eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CG101 high dose (Experimental): Patient in this group received high dose CG101 eyedrops in period 1 (0W to 4W) and received placebo in period 2 (8W to 12W).
  Interventions: Drug: CG101 high dose + artificial tear; Drug: placebo + artificial tear
- CG101 low dose (Experimental): Patient in this group received low dose CG101 eyedrops in period 1 ( 0W to 4W) and received high dose CG101 eyedrops in period 2 ( 8W to 12W).
  Interventions: Drug: CG101 high dose + artificial tear; Drug: CG101 low dose + artificial tear
- Placebo (Placebo Comparator): Patient in this group received placebo eyedrops in period 1 (0W to 4W) and received low dose CG101 eyedrops in period 2 (8W to 12W).
  Interventions: Drug: CG101 low dose + artificial tear; Drug: placebo + artificial tear

INTERVENTIONS:
Drug: CG101 high dose + artificial tear — Patient in this group received high dose CG101 eyedrops twice daily and artificial tear three times a day during week 0 to week 4, after 4 week washout, patient in this group cross over to receive placebo CG101 eyedrops twice daily and artificial tear three times a day during week 8 to week 12.
  Other Names: 2-3
  Arms: CG101 high dose; CG101 low dose
Drug: CG101 low dose + artificial tear — Patient in this group received low dose CG101 eyedrops twice daily and artificial tear three times a day during week 0 to week 4, after 4 week washout, patient in this group cross over to receive high dose CG101 eyedrops twice daily and artificial tear three times a day during week 8 to week 12.
  Other Names: 1-2
  Arms: CG101 low dose; Placebo
Drug: placebo + artificial tear — Patient in this group received placebo dose CG101 eyedrops twice daily and artificial tear three times a day during week 0 to week 4, after 4 week washout, patient in this group cross over to receive low dose CG101 eyedrops twice daily and artificial tear three times a day during week 8 to week 12.
  Other Names: 3-1
  Arms: CG101 high dose; Placebo

SUMMARY:
This study is a single-center, randomized, double-blind, placebo-controlled, cross-over clinical trial designed to evaluate the effectiveness and safety of CG-101 eye drops for the treatment of dry eye syndrome, using a placebo as a control.

DETAILED DESCRIPTION:
This study is a single-center, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the effectiveness and safety of CG-101 eye drops for the treatment of dry eye syndrome, using a placebo as a control. The treatment period lasts for 84 days. Participants are randomly assigned to in randomized sequence.

There are three sequence, including sequence 1 (CG101 high dose in period 1 switch to placebo in period 2), sequence 2 (CG101 low dose in period 1 swich to CG101 high dose in period 2), and sequence 3 (placebo in period 1 swithc to CG101 high dose in period 2). Period 1 starts from 0W to 4W, then washout period lasts from 4W to 8W, and period 2 starts from 8W to 12W. Participant will need to visit the clinic at 2W, 4W 8W, 10W, 12W after enrollment for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all the following inclusion criteria to be enrolled in this study:

1. Age ≥ 18 years, regardless of gender;
2. Clearly understand and voluntarily participate in the study, with the ability and willingness to sign a written informed consent form (ICF) and comply with all study assessments and visits as instructed;
3. Male and female participants of childbearing potential must agree to use medically acceptable contraception during the study and for 3 months (90 days) after the study ends. Women who are not postmenopausal or have not been menopausal for less than two years (from the last menstrual period to the signing of the ICF) must have a negative pregnancy test at Visits 0 and 1.
4. A history of bilateral dry eye disease prior to the screening visit (i.e., at least one of the following subjective symptoms: ocular dryness, foreign body sensation, burning sensation, fatigue, discomfort, redness, or fluctuating vision);
5. Recent use (within 30 days prior to Visit 0) of artificial tears to relieve dry eye symptoms, with discontinuation of artificial tears at least 72 hours before Visit 0;
6. Ocular Surface Disease Index (OSDI) total score ≥ 13 at Visit 0;
7. Best corrected visual acuity ≥ 4.3 (5-point recording method on the international standard logarithmic visual acuity chart at 5 meters) in both eyes at Visit 0;
8. At least one eye must have a positive corneal fluorescein staining score (CFS) at Visits 0 and 1;
9. Non-anesthetic tear secretion test (SIT) ≤ 10 mm/5 min at Visits 0 and 1;
10. Tear film break-up time (BUT) ≤ 10 seconds at Visits 0 and 1.

Exclusion Criteria:

* **Medical History**

  1. History of malignant tumors in or around the eyes;
  2. Dry eye formed due to scarring (e.g., radiation, alkali burns, Stevens-Johnson syndrome, scarring pemphigoid) or destruction of conjunctival goblet cells (e.g., vitamin A deficiency);
  3. Active ocular allergy or a history of possible ocular allergy during the study period;
  4. Presence of ocular or systemic infection (bacterial, viral, or fungal) at Visits 0 and 1, including fever and herpetic keratitis, or currently receiving antibiotic treatment;
  5. History of glaucoma diagnosis;
  6. History of any immunodeficiency, HIV infection, hepatitis B or C, acute active hepatitis (anti-HAV IgM positive), organ or bone marrow transplantation;
  7. Presence of any significant chronic diseases that the investigator considers may interfere with study parameters, including but not limited to: severe pulmonary diseases, poorly controlled hypertension, and/or poorly controlled diabetes;
  8. Blood donation or significant blood loss (more than 400 ml) within 56 days before Visit 0;

     **Physical or Laboratory Examination Abnormalities**
  9. Presence of active rosacea-related ocular lesions, periorbital acne, or pterygium in the eyes or eyelids;
  10. Anatomical abnormalities of the eyelids (e.g., eyelid laxity, entropion, or ectropion) or abnormal blinking patterns;
  11. Abnormal findings during slit-lamp and/or fundus examination during the screening period, which the investigator deems clinically significant (including but not limited to conjunctivitis, trichiasis, conjunctival laxity, glaucoma, uveitis), requiring pharmacological treatment and believed by the investigator to potentially interfere with trial results;

      **Previous Medications and Treatments**
  12. Intraocular surgery or ocular laser surgery, YAG laser capsulotomy, or any surgery affecting the meibomian glands within the 180 days prior to Visit 0, or plans to undergo such surgery or treatment during the study;
  13. Punctal occlusion or surgical removal of plugs (resorbable plugs within 180 days) within 60 days before Visit 0, or plans to undergo punctal occlusion or surgical removal of plugs during the study;
  14. Use of systemic immunomodulators, oral doxycycline or tetracycline within 90 days before Visit 0, or plans to use these medications irregularly during the study;
  15. Local use of immunomodulators (e.g., cyclosporine A eye drops, tacrolimus eye drops) within 30 days before Visit 0;
  16. Use of any medications known to cause dryness of the eyes (e.g., diuretics, antidepressants, decongestants, antispasmodics, antihistamines, anesthetics, etc.) within 30 days before Visit 0, or plans to use these medications irregularly during the study;
  17. Active blepharitis or meibomian gland dysfunction and treatment for the eyes (e.g., eyelid scrubs, meibomian gland massage, wet compresses, hot compresses, systemic antibiotics, and other oral medications for ocular disease) within 30 days before Visit 0, or plans to treat irregularly during the study;
  18. Use of corticosteroids or mast cell stabilizers (including ocular) within 30 days before Visit 0;
  19. Use of contact lenses within 14 days before Visit 0, or plans to continue using them during the study;
  20. Known allergies to test drugs or their excipients, fluorescein, or other substances involved in examination;

      **Other**
  21. Pregnant, nursing, or planning to become pregnant;
  22. A family member residing in the same household has already been enrolled in this study or is a direct relative of staff directly involved in the management or support of this study;
  23. Undergoing a drug or device trial within 30 days or 5 half-lives (whichever is longer) prior to screening, judged by the investigator to potentially affect trial results, or during the study may necessitate participation in other drug or device trials;
  24. Situations that the investigator/sponsor believes may expose participants to significant risk, potentially confound trial results, seriously interfere with a participant's ability to participate in the study (e.g., language barriers, illiteracy), or not be in the best interest of the participant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-05-22 (Estimated); Study Completion 2025-05-22 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Corneal Staining Scores at Week 4 | Baseline, Week 4
  Corneal staining was assessed using fluorescein dye, a yellow filter, and a slit lamp. The cornea was divided into 5 different zones. Each corneal zone was graded independently using a 0 to 3 grading scale; where 0=none, 1=slight, 2=moderate, 3=severe. Sum of scores of each zone led to total score. Total score range: 0 to 15, higher score indicated greater staining. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.
Percentage of Participants With Systemic Adverse Events (AEs) | Baseline up to Week 12
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Systemic AEs are the events which are not localized but occur throughout the systemic circulation.
Percentage of Participants With Ocular Adverse Events (AEs) | Baseline up to Week 12
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Ocular AEs are the events which are localized in the ocular region.
Percentage of Participants With Ocular Tolerability Assessment | Baseline up to Week 12
  Ocular tolerability assessment included evaluation of severity and duration of the 5 symptoms: burning/stinging, blurred vision, ocular discomfort, pain, tearing. Severity was assessed on a 4-point scale, where 0=none, 1=mild, 2=moderate and 3=severe. Duration was assessed as immediate (if subsided within 5 minutes [<5 min] after application) or persistent (if continued beyond 5 minutes [>=5 min] after application).
Change From Baseline in Tear Break-up Time (TBUT) at Week 4 | Baseline, Week 4
  TBUT was the time interval between the last complete blink and the first appearance of a dry spot, or disruption in the tear film. It was measured under a slit lamp following instillation of fluorescein dye in the eye using a stopwatch. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline
Change From Baseline in Ocular Surface Disease Index (OSDI) Total and Subscale Score at Week 4 | Baseline, Week 4
  OSDI is a validated instrument for ocular surface disease. It has 12 items, each measured on 5-point Likert scale (0=none of the time, 4=all the time). Based on these item scores, a total OSDI score (question 1 [Q1]-Q12) and three subscale scores can be derived: Ocular Symptom (Q1-Q3), Vision-related function (Q4-Q9), and Environmental trigger (Q10-Q12). Each derived score ranges from 0 to 100, with a higher score indicates worse condition.
Change From Baseline in Schirmer Wetting Score With Anesthesiaout at Week 4 | Baseline, Week 4
  Schirmer test without anesthesia: well standardized test used to estimate tear flow stimulated reflexly by insertion of a filter paper strip into the conjunctival sac for 5 min. The length of wetting was recorded to the nearest 0.5 mm. If the wetting line was oblique, halfway point was used. Results from study eye are reported. Study eye is the 'worse eye', defined as the eye with worse Schirmer test score without anesthesia score at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol